CLINICAL TRIAL: NCT07176195
Title: The Impact of Eating Habits on the Health of Employees in the Defense Sector
Acronym: PRENAV
Status: Active, not recruiting | Type: Observational
Sponsor: University of Primorska (Other)
Collaborators: University of Ljubljana, Faculty of Social Sciences (Unknown); Ministry of Defence, Slovenia (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Assoc. Prof. Dr., University of Primorska
Other Study IDs: PRENAV
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood for biochemical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PRENAV project focuses on healthy and sustainable eating among employees in the defense sector of the Republic of Slovenia. The project pursues two main objectives:

1. In a selected sample of employees in the defense sector, the project will determine their nutritional status and assess indicators of metabolic health, including serum concentration of vitamin D.
2. In the selected sample, through a survey and qualitative methods (interviews, focus groups), we will identify the eating habits of employees in the defense sector, the factors influencing their dietary decisions, and the barriers and facilitators of healthy and sustainable eating among employees in the defense sector.

Based on these findings, we will prepare recommendations and an action plan to promote healthier and more sustainable eating among employees in the defense sector.

DETAILED DESCRIPTION:
Participants will be selected using non-probability quota sampling, with quotas defined according to population characteristics, taking into account the research problem:

1. Proportional representation based on the permanent composition of employees in the defense sector: soldiers, non-commissioned officers, officers, and military staff (military personnel 70%) and civilian employees (30%).
2. Eating habits (canteens) during working hours: based on the number of employees at each military barracks (n=13) and at the Ministry of Defence.
3. Gender structure of the observed population: military personnel 85% male and 15% female; civilian employees according to the gender distribution data of the civilian workforce.
4. The purpose of this sampling strategy is to proportionally capture those characteristics of the military and civilian population employed in the defense sector that are crucial for the research objectives, namely: employment structure, gender distribution, and eating habits in canteens.

ELIGIBILITY:
Inclusion Criteria:

* Adults employed at the Ministry of Defence or in the military.
* Asymptomatic individuals (i.e., without current acute illness or relevant health complaints).
* Willingness to provide informed consent to participate in the study.
* Willingness and ability to complete all questions in the Food Frequency Questionnaire (FFQ) and other study questionnaires.

Exclusion Criteria:

* Pregnant and breastfeeding women, as well as individuals with electronic implants such as a pacemaker, will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be adults, with an expected age range of 18-65 years, including both males and females, employed in the defense sector. Participants will include both military personnel and civilians.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Food intake | From enrollment to the end of the November 2025
  Participants of the cross-sectional study will complete a Food Frequency Questionnaire (FFQ), adapted for the Slovenian population (Bizjak, Jenko Pražnikar & Koroušić Seljak, 2014), with the aid of visual materials (portion size images). In the FFQ method, respondents answer questions about the frequency of consumption of specific foods over a certain period of time.
  From a methodological perspective, most studies examining dietary habits and food/nutrient intake in military populations use the Food Frequency Questionnaire (FFQ), which is typically adapted to the general population of individual countries (Collins et al., 2021), rather than specifically tailored to the military population.
  The questionnaire is based on self-reporting by study participants. It is an internationally established methodology for subjective assessment of nutrient intake, and the risk for participants is negligible.

SECONDARY OUTCOMES:
Body muscle mass (kg) | From enrollment to the end of November 2025
  Body composition will be analyzed using the BodyStat1500 body analyzer. Bioelectrical impedance measurements will be conducted according to the standard protocol recommended by the European Society for Clinical Nutrition (Kyle et al., 2004). The protocol specifies that measurements should be taken on an empty stomach, with an emptied bladder, without physical activity or alcohol intake in the past 8 hours.
  Participants will lie in a supine position for at least 5-10 minutes before the measurement, following the standard protocol (we will use 10 minutes in the supine position). Electrodes will be placed tetrapolarly on cleaned skin: on the right arm (from fingers to wrist) and the leg (instep to ankle). The distance between the two electrodes must be at least 5 centimeters. The participants' arms will be positioned at a 30-degree angle relative to the torso, and the legs spread at a 45-degree angle.
vitamin D (ng/ml) | From enrollment to the end of the November 2025
  Serum levels of vitamin D will be measured in biochemical laboratory of General Hospital of Izola, Slovenia.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - University of Primorska Faculty of Health Sciences, Izola, Izola
  - University of Ljubljana Faculty of Social Sciences, Ljubljana, Ljubljana